CLINICAL TRIAL: NCT05553444
Title: The Effect of a Self-management Intervention on Pain Intensity and Functional Disability in Adolescent Patients With Low Back Pain - a Single Case Experimental Study.
Brief Title: Effect of Self-management Intervention on Pain Intensity and Functional Disability in Adolescent Patients With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Christian Lund Straszek, M.Sc. Ph.D Fellow, Aalborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAM-AAU 241-2
Record Dates: First submitted 2022-08-24; First posted 2022-09-23 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Single subject experimental design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self-management intervention (Experimental): The intervention is based on the 5 key skills for successful self-management which are;
  1. Problem solving
  2. Decision-making
  3. Utilizing resources
  4. Forming partnerships with healthcare providers
  5. Taking action. It is important to keep in mind, that not all included patients will necessarily lack all 5 skills. As such, the intervention will be tailored to each participant based on the initial assessment and continuous clinical reasoning.
  Interventions: Behavioral: Self-management intervention

INTERVENTIONS:
Behavioral: Self-management intervention — The procedure will be based on the A - B - A'/B' design. After recruitment, patients will attend an initial session with CLS where written and oral information about the study will be provided. In this study, the A phase will serve as baseline to establish fluctuation in pain intensity prior to initiating the treatment.
  During phase A, patients will be assessed every day for a minimum of 8 days and maximum of 14 days.
  During phase B, CLS will facilitate the intervention based on the initial session, pain levels during phase A and the patients' goals. During phase B, patients will attend a 1-hour weekly session over 6 weeks.
  During phase A', the participants will be followed weekly for 12 weeks. During the phase A', participants will not receive treatment.
  Phase B' contains 3 x 1 hour criterion-based booster sessions which are delivered over 3 consecutive weeks.

SUMMARY:
Low back pain (LBP) is prevalent among adolescents from the general population and in general practice. Not only is LBP associated with pain and functional limitation among patients, also the socioeconomic burden of the condition is substantial worldwide. Chronic cases of LBP are not uncommon in adolescents, especially among those whose parents are suffering from chronic pain. Several individual factors influence LBP among adolescents. Especially previous episodes of LBP, low pain self-efficacy levels and worries about LBP has been identified as worsening factors in regard to pain and disability.

At present there is little evidence to inform a large randomized experimental study to investigate the effect of a given treatment modality in this group of young patients. Furthermore, it remains to be investigated if individual factors, such as, pain self-efficacy levels and worries about LBP may mediate the effect of a behavioral intervention regarding pain and disability. However, the single case experimental design allows for close monitoring of the patients during a controlled treatment course. As such, the single case experimental design study can provide vital and fundamental knowledge regarding treatment effect and mediating factors in relation to an intervention aimed at improving self-management in adolescent LBP patients.

This study aims to investigate the effect of an intervention to improve self-management among adolescent LBP patients assessed by pain intensity and functional disability in a single case experimental design. We further aimed to investigate if LBP related worries and pain self-efficacy would mediate the effect of the intervention. We hypothesized that the self-management intervention would lead to lower pain intensity scores and decrease disability levels on a patient level.

ELIGIBILITY:
Inclusion Criteria:

1. 15-19 years of age.
2. Experience consistent or fluctuating axial LBP (between T12 and the gluteal fold) for more than 30 days prior to inclusion.
3. Worst pain intensity during the past 24 hours equal to or more than 3 on 0-10 Numeric Pain Rating Scale (NPRS).

Eligible patients are also required to meet two of the following three criteria:

1. Experience functional limitations in one or more daily activities (e.g. sports participation, sitting or lifting). Functional limitation will be assessed with the Patient Specific Functional Scale (PSFS). Patients is characterized as experiencing functional limitations if they score 8 or below on an 11-point scale (0, unable to perform activity; 10, able to perform activity at pre-injury level) in regards to one self-reported activity.
2. Being absent from work and/or school for one or more days during the past 30 days due to LBP.
3. Being worried about their back pain (i.e. scoring 3 or higher on a 0-10 scale in relation to the question; "Are you worried about your back pain" - see the Illness perception item described below).

Exclusion Criteria:

Participant are excluded if they are diagnosed with rheumatic arthritis or a primary neurological disorder (e.g. multiple sclerosis), have an underlying pathology such as infection, cancer or fracture or shows clinical symptoms of cauda equina.

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Functional limitations | Will be assessed throughout the study. The primary outcome will be functional limitations 20 weeks after inclusion.
  In this questionnaire, the participants will identify one to three activities which they find themselves limited accomplishing. These activities are rated from a 0 (unable to perform activity) to 10 (able to perform activity at pre-injury level). The primary outcome for each patient will be the activity with the lowest score on the PSFS. If two or more activity have equally low scores, the patient will determine which should be the primary outcome
Self-reported pain intensity | Will be assessed throughout the study. The primary outcome will be pain intensity 20 weeks after inclusion.
  The 11-point Numeric Pain Rating Scale (NRPS) (0 equals no pain and 10 equals worst possible pain) will be used to assess worst pain during the past 24 hours.

SECONDARY OUTCOMES:
Pain Self-efficacy | Assessed at baseline (T0), after 8-14 days (T1), after addtional 6 weeks (T2) and after addtional 12 weeks (T3)
  Will be assess with the 2-item short form of the Pain Self-Efficacy Questionnaire. This questionnaire is based on 2 items evaluating to which degree patients feel confident in engaging in different task despite pain being present. Each question has a corresponding 7-point Likert scale ranging from 0 (not confident at all) to 6 (very confident).
Pain interference | Assessed at baseline (T0), after 8-14 days (T1), after addtional 6 weeks (T2) and after addtional 12 weeks (T3)
  Please check the box which best describes how your back pain affects your usual activities through a normal day (e.g. go to school, participate in sport, be with friends and family". This question will have the following 5 response options.

OTHER OUTCOMES:
Ilness perception | Assessed at baseline (T0), after 8-14 days (T1), after addtional 6 weeks (T2) and after addtional 12 weeks (T3)
  "Are you worried about your back pain"? The response options will be a 11-point scale with 0 being equal to "not worried at all" whereas 10 will be equal to "very worried"
Physical activity | Assessed at baseline (T0), after 8-14 days (T1), after addtional 6 weeks (T2) and after addtional 12 weeks (T3)
  "How often do you usually exercise at a level where you get short of breath or sweat". This question will have 7 response options.
Health-related quality of life | Assessed at baseline (T0), after 8-14 days (T1), after addtional 6 weeks (T2) and after addtional 12 weeks (T3)
  Will be assessed with two questions:
  "Have you felt satisfied with your life?" The response options for this question are; not at all, slightly, moderately, very and extremely
  "Have you felt under pressure?" The response options for this question are; never, seldom, quite often, very often, always.
The Global Rating of Change | Assessed after 6 weeks (T2) and after addtional 12 weeks (T3)
  The Global Rating of Change Scale (GROC) will be used to assess self-reported improvement. The scale is based on a single question along with a 7-point Likert scale ranging from "much improved" to "much worse".
Patient Acceptable Symptom State | Assessed after 6 weeks (T2) and after addtional 12 weeks (T3)
  The Patient Acceptable Symptom State (PASS) consists of a single question; "Who do you experience you LBP now compared to before you initiated the treatment", with a yes/no response option.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for General Practice at Aalborg University, Aalborg, Northern Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No